CLINICAL TRIAL: NCT01051089
Title: Effects of Lifestyle Modification Focusing on Exercise Intervention on Risk of Atherosclerosis and Metabolic Parameters in Type 2 Diabetic Patients
Brief Title: Effects of Lifestyle Modification on Metabolic Parameters in Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Moonsuk Nam, MD, PhD, Inha University School of Medicine, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-459
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; lifestyle modification
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Lifestyle modification (Experimental): supervised exercise with diet education
  Interventions: Behavioral: Lifestyle modification
- Control (No Intervention): Control (ordinary care with usual education)

INTERVENTIONS:
Behavioral: Lifestyle modification — Exercise and diet education
  Arms: Lifestyle modification

SUMMARY:
The study is a randomized controlled study comparing the metabolic effect of a 3 month intensive lifestyle modification intervention in Korean type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* age 25 or older,
* type 2 diabetes mellitus,
* HbA1c 6.5-10% BMI 23 or higher.

Exclusion Criteria:

* type 1 diabetes,
* recent (within 3 months) cardiovascular event,
* severe hepatic or renal dysfunction,
* insulin use,
* glucocorticoid use.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c, serum adipokine levels | 3 months

SECONDARY OUTCOMES:
Body composition | 3 months
Pulse wave velocity | 3 months
Insulin secretion and sensitivity | 3 months
VO2max | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea